CLINICAL TRIAL: NCT05572281
Title: An Open-Label, Two-Period, Randomized, Single Oral Dose, Crossover Study to Evaluate the Bioequivalence of Tasimelteon Capsule Formulation Relative to Tasimelteon Liquid Suspension Formulation in Healthy Volunteers
Brief Title: Bioequivalence Study Between Tasimelteon Capsule Formulation and Liquid Suspension Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VP-VEC-162-1113
Record Dates: First submitted 2022-07-05; First posted 2022-10-07 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — tasimelteon

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): tasimelteon liquid suspension formulation then tasimelteon capsule formulation
  Interventions: Drug: Tasimelteon Oral Capsule; Drug: Tasimelteon Oral Suspension
- Sequence B (Experimental): tasimelteon capsule formulation then tasimelteon liquid suspension formulation
  Interventions: Drug: Tasimelteon Oral Capsule; Drug: Tasimelteon Oral Suspension

INTERVENTIONS:
Drug: Tasimelteon Oral Capsule — No additional information
Drug: Tasimelteon Oral Suspension — No additional information

SUMMARY:
This is a single center, two-period, randomized study to evaluate the bioequivalence of a single dose of tasimelteon capsule formulation relative to a single dose of liquid suspension formation in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female participants between 18 to 55 years (inclusive).
* Good health as determined by no clinically significant deviations from normal in medical history, clinical laboratory determination, ECGs, and physical examinations conducted during the screening visit.
* Participants with no clinically significant medical, psychiatric or sleep disorders as determined by the PI.

Exclusion Criteria:

* Participants with history of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Participants who suffered from significant physical illness (required hospitalization) in the 4-week period preceding baseline will be excluded.
* Participants with history of smoking or use of tobacco products in the last 3 months.
* Pregnant or nursing (lactating) women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Bioequivalence between tasimelteon capsule formulation relative to tasimelteon liquid suspension formulation | 8 hours
  as measured by plasma concentrations
Assessment of Safety and Tolerability of the liquid suspension and capsule formulation of tasimelteon | 7 days
  as measured by incidence of adverse events and clinically significant changes in laboratory values, ECG parameters, and vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No